CLINICAL TRIAL: NCT03542188
Title: TReatment Strategy In Acute Ischemic larGE Vessel STROKE: Prioritize Thrombolysis or Endovascular Treatment
Acronym: TRIAGE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Aarhus (Other)
Collaborators: Aarhus University Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CT1-10-72-28-18
Record Dates: First submitted 2018-05-16; First posted 2018-05-31 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-12

CONDITIONS: Stroke
Keywords: Large Vessel Occlusion; Stroke; EVT
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Who Masked: Investigator
Masking Description: Single-blinded
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Primary Stroke Center (PSC) (Active Comparator): Transport to a primary stroke center for early IV-thrombolysis followed by a secondary transport to a comprehensive stroke center for EVT if needed.
  Interventions: Behavioral: Primary Stroke Center (PSC); Behavioral: Comprehensive Stroke Center (CSC)
- Comprehensive Stroke Center (CSC) (Experimental): Direct transport to a comprehensive stroke center for IV-trombolysis and early EVT.
  Interventions: Behavioral: Comprehensive Stroke Center (CSC)

INTERVENTIONS:
Behavioral: Primary Stroke Center (PSC) — Transport to a primary stroke center for early IV-thrombolysis followed by a secondary transport to a comprehensive stroke center for EVT if needed.
  Arms: Primary Stroke Center (PSC)
Behavioral: Comprehensive Stroke Center (CSC) — Direct transport to a comprehensive stroke center for IV-thrombolysis and early EVT.

SUMMARY:
Should we prioritize thrombectomy or thrombolysis in acute stroke? Finding the answer to this question will improve treatment and outcome for stroke patients only by changing triage and transportation. And it will have implications for stroke patients around the world.

The investigators propose a national investigator-driven, multi-center, randomised single-blinded clinical trial to investigate which treatment strategy is superior in patients with acute stroke and suspected large vessel occlusion (LVO): direct transport to a comprehensive stroke center for early endovascular therapy (EVT) or to a primary stroke center for early IV thrombolysis followed by secondary transport to a comprehensive stroke center for EVT if needed.

Effective reperfusion therapy marks a new era within stroke medicine and has been driving major changes in the organization of care within the last decade. Timely thrombolysis and/or EVT in acute ischemic stroke is a key factor for improved outcome. Major stroke occur in 25% of all cases and is caused by LVO. Major strokes have approximately 60% risk of severe disability or death at three months if not treated. EVT is superior to thrombolysis in strokes caused by a LVO, but EVT is only performed in specialized centers due to the complexity of the treatment and need for skilled neurointerventionalists.

A simple stroke severity score has been developed, that can identify most patients with LVO in the pre-hospital setting. This enables selection of patients with a suspected LVO to be transported without delay directly to a comprehensive stroke center for EVT while potentially bypassing a nearer primary stroke center for IV-thrombolysis.

Study results will have major impact of future acute stroke treatment and organization.

DETAILED DESCRIPTION:
Project description In the new area of reperfusion therapy for acute ischemic stroke (AIS) a major question has emerged: Should the Emergency Medical Service take the patient to the nearest primary stroke center (for fast thrombolysis) or should they bypass the primary stroke center and take the patient directly to a comprehensive stroke center with endovascular capabilities? We propose a randomized controlled single-blind trial to explore this worldwide clinical dilemma.

Objective To determine if direct transport to a comprehensive stroke center improves outcome for patients with suspected large vessel occlusion (LVO) that occur in the catchment area of a primary stroke center without potentially harming patients who only need thrombolysis.

Hypothesis

The guidelines tell us to admit a stroke patient to the nearest stroke hospital. The investigators wish to perform the study because we believe that in case of LVO, direct transport to a comprehensive stroke center is a better strategy. The investigators hypothesize that:

* A symptom based triage strategy in the catchment area of the primary stroke center results in net benefit for patients with AIS.
* AIS patients with a LVO occurring in a primary stroke center catchment area will have better clinical outcome at 90 days if they are transported directly to a comprehensive stroke center.
* AIS patients without LVO at admission might be subjected to a longer transport to a comprehensive stroke center and a longer delay to IV thrombolysis, but this will not translate into a poorer prognosis for patients with AIS.
* Patients suspected to have LVO who turn out to have ICH or stroke mimics after imaging on admission will not be harmed from being randomized to alternative pre-hospital transport strategies.

The investigators formulate the null hypothesis:

The transport strategy of an ischemic stroke patients does not influence outcome.

Review of existing knowledge in the field The possibility of effective reperfusion therapy marks a new era within treatment of stroke and has been driving major changes in the organization of care within the last decade. Timely IV-thrombolysis and/or endovascular therapy (EVT) in acute ischemic stroke is a key factor for improved outcome. Major stroke occur in 25% of all cases and is caused by large vessel occlusion (LVO). Major strokes have approximately 60% risk of severe disability or death at three months if not treated. EVT is superior to IV-thrombolysis in strokes caused by a LVO (1), but not every IV-thrombolysis center can perform endovascular therapy due to the complexity of the treatment and need for skilled neurointerventionalists.

Methods and materials A national investigator-driven, multi-center, randomized, single-blinded, clinical trial to investigate which logistic strategy is best in acute stroke with suspected LVO: direct transport to a comprehensive stroke center for early EVT or to a primary stroke center for early IV-thrombolysis followed by a secondary transport to a comprehensive stroke center for EVT if needed (TRIAGE-STROKE).

Prehospital identification of LVO The patient with a suspected LVO is the focus of our study. At the same time, the investigators do not wish to "harm" the patients without a LVO by giving them a longer time to treatment.

The patient or a bystander will have called for help and the Emergency Medical Service will be send to the patient. To identify LVO the investigators will use the PASS scale in the prehospital examination: The patient is asked the month and age, gaze palsy and/or deviation is registered and arm drift is examined. A score of 2 or 3 points at PASS predict a LVO. PASS is implemented i a new score system called Prehospital Stroke Score (PreSS) as PreSS part 2 in the central region of Denmark.

If the "pick up" place is near a comprehensive stroke center, the patient will be admitted there regardless of the score. If the "pick up" place is nearer a primary stroke center, the patient will enter STROKE-TRIAGE. In both cases admission is agreed after telephone contact between ambulance and the senior "EVT/thrombolysis doctor" on call. At admission whether at the primary or the comprehensive stroke center indication for IV thrombolysis and EVT treatment will be evaluated according to national clinical guidelines for IV thrombolysis/EVT treatment.

Randomization and consent The investigators will conduct the study as an acute study and randomize between the two transport strategies without consent, as it is not possible to obtain consent from patient or relative prior to randomization. The patients and their relatives will be informed afterwards that the patient was enrolled in a study, but that the study only involved the transport strategy and that they otherwise received standard treatment We will ask for his acceptance to be in the study to collect his or her medical information for research purposes. The patient can withdraw consent anytime.

The patient will be randomized for primary transport to either the primary stroke center or the comprehensive stroke center. The randomization will be 1:1.

Data collection and statistics Follow-up of all patients with suspected stroke is possible by unambiguous individual level record linkage between high quality nationwide population-based registries using the unique individual civil registration number (CPR), which is provided to all Danish citizens upon birth or immigration. For patients with a confirmed stroke diagnosis after in-hospital diagnostic work-up the investigators will collect all pre-hospital time registrations, all demographic and stroke related data from the Danish Stroke Register and electronic prehospital patient records located at the regional Emergency Medical Communication Centers.

Baseline characteristics will be summarized by means of simple descriptive statistics. The primary analysis consists of a comparison of the primary outcome after 90 days between the trial treatment groups. In all analyses, statistical precision will be expressed by means of 95% CI. A detailed statistical analysis plan will be prepared prior to the start of analyses.

Risks and Safety It sounds reasonable that patients with LVO might benefit from faster transport to a comprehensive stroke center, but by subjecting a group of stroke patients to a longer transport, patients who at admission only need IV-thrombolysis or have intracerebral hemorrhage (ICH), will risk a longer time to their treatment. This may happen in a small number of AIS patients with spontaneous clot resolution during transport or the clot may be too distal to be reached by catheter. The balance of risk versus benefit of the two logistic approaches is unknown. For patients where imaging at admission show an ICH a longer transport time is not known to expose the patient to any harm.

If the local investigator or other member of the team at a center have a concern about the outcome of their trial procedures, they should inform the trial coordinator, which will organize a blinded assessment of the relevant outcome events

Ethical considerations Since the majority of the patients are incompetent at admission and since the treatment is severely time dependent, the investigators find that the conditions for an acute study are fulfilled. Eventually some patients randomized in the ambulance have an ICH or stroke mimic i.e. tumor. These patients will not be exposed to any harm from a potential longer transport time, since treatment is not severely time dependent. Furthermore, ICH patients may profit if transported directly to a comprehensive stroke center easy access to neurosurgery service.

Lastly, there is equipoise as to what transport strategy is best, so the patients will not risk getting a lower-than standard treatment.

The clinical study will be conducted, and essential documentation archived, in compliance with UCR SOPs and standards, which incorporate the requirements of the ICH Guideline for Good Clinical Practice and EN ISO 14155:2011(E).

Cost-effectiveness analysis A full cost-effectiveness analysis will be conducted according to international guidelines for the economic evaluation alongside clinical trials. Patient specific data for resource usage will be retrieved from Danish registries (covering the period from one year prior to one year after enrolment), and a micro costing study will be conducted to estimate the extra time and resources at the clinics needed to bypass the PSC for patients with symptoms of large- vessel occlusion compared to usual practice. A full health economic evaluation including a budget impact analysis will be conducted to illustrate the incremental costs and gained QALYs as well as the total national costs and consequences of bypassing the PSC for same patient group nationwide in Denmark.

Sample size Based upon previous trials the investigators have estimated that a good outcome can be measured by including a little less than 300 patients in each arm. We aim at including 600 patients. Samplesize is reestimated as soon as 200 patients have been followed up

ELIGIBILITY:
Inclusion Criteria:

1. Symptoms of acute stroke
2. No contraindication for IV thrombolysis
3. Stroke occurring ("pick up" place) in catchment area of a primary stroke center
4. The patient has Pre-hospital Acute Stroke Severity (PASS) score ≥2
5. Pre-stroke modified Rankin Score 0-2 (meaning living independently.)
6. Feasible to start IV-thrombolysis within 4.5 hours at CSC

Exclusion Criteria:

1. Syncope
2. Seizure
3. Known diagnosis of epilepsy
4. Medical condition and no signs of stroke (e.g. hypoglycemia)
5. In-hospital strokes
6. Life expectancy of less than 1 year.

Exclusion criteria for the analysis of the ischemic patients (to be determined after admission at stroke center)

1. Imaging showing ICH
2. Stroke mimics

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 174 (Actual)
Dates: Start 2018-09-03 (Actual); Primary Completion 2022-08-31 (Actual); Study Completion 2022-08-31 (Actual)

PRIMARY OUTCOMES:
mRS score after 90 days for AIS patients | 90 days
  Blinded outcome of functional disability at 90 days using modified Rankin Score (mRS) ranging from no symptoms (score 0) to dead (score 6) analyzed as shift analysis in all patients ending with diagnosis of AIS.

SECONDARY OUTCOMES:
mRS score after 90 days (shift analysis) for all randomized. | 90 days
  Blinded outcome of functional disability at 90 days using modified Rankin Score (mRS) ranging from no symptoms (score 0) to dead (score 6) analyzed as shift analysis in all randomized patients
mRS score after 90 days (shift analysis) for AIS patients without LVO | 90 days
  Blinded outcome of functional disability at 90 days using modified Rankin Score (mRS) ranging from no symptoms (score 0) to dead (score 6) analyzed as shift analysis in all patiens without LVO
mRS score after 90 days (shift analysis) for patients with hemorrhagic stroke | 90 days
  Blinded outcome of functional disability at 90 days using modified Rankin Score (mRS) ranging from no symptoms (score 0) to dead (score 6) analyzed as shift analysis in all with hemorrhagic stroke
mRS score after 90 days (shift analysis) for patients with stroke mimics | 90 days
  Blinded outcome of functional disability at 90 days using modified Rankin Score (mRS) ranging from no symptoms (score 0) to dead (score 6) analyzed as shift analysis in all patients with stroke mimics
mRS score ≤2 (independent) after 90 days for AIS patients treated with EVT | 90 days
  Blinded outcome of functional disability at 90 days using modified Rankin Score (mRS) ranging from no symptoms (score 0) to dead (score 6) analyzed as shift analysis in all patients treated with EVT
Severe dependency or death after 90 days for AIS patients treated with EVT | 90 days
  mRS score 5+6 (severe dependency or death) after 90 days for AIS patients treated with EVT. (Safety endpoint.)
Severe dependency or death after 90 days in patients with hemorrhagic stroke | 90 days
  mRS score 5+6 (severe dependency or death) after 90 days in patients with hemorrhagic stroke. (Safety endpoint.)
Times (from onset, pick-up and arrival) to groin puncture for patients treated with EVT | 1 day
  Mean time to groin puncture for patients treated with EVT
Times (from onset, pick-up and arrival)to IV thrombolysis for patients treated with IV thrombolysis only. | 1 day
  Mean time to IV thrombolysis for patients treated with IV thrombolysis only. (Safety endpoint.)
Successful re-perfusion in EVT treated | 1 day
  modified Trombolysis In Cerebral Iscemia (TICI) 2b-3
Length of stay at CSC for all patients withpot LVO | 1 week
  Median time in hours at CSC

OTHER OUTCOMES:
TimesEVT | up to 24 hours
  (from onset, pick-up and arrival) to groin puncture for patients treated with EVT (Mean time to groin puncture for patients treated with EVT)
TimesIVT | up to 24 hours
  (from onset, pick-up and arrival) to IV thrombolysis for patients treated with IV thrombolysis only. Time to IV thrombolysis for patients treated with IV thrombolysis only (bypass vs. direct transport.) (Safety endpoint.)
Successful reperfusion | up to 24 hours
  modified Thrombolysis In Cerebral Ischemia 2b-3) in EVT treated (bypass vs. direct transport
Length of stay at CSC | up to 30 days
  Length of stay at CSC for all patients without LVO
QUALY | up to 4 months
  Quality of life qual-5

CONTACTS AND LOCATIONS:
Overall Officials: Claus Z Simonsen, MD, PhD, Principal Investigator — Aarhus University Hospital; Grethe Andersen, Professor, Study Director — Aarhus University Hospital
Locations (1):
- Aarhus University Hospital, Aarhus, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Southerland AM, Johnston KC, Molina CA, Selim MH, Kamal N, Goyal M. Suspected Large Vessel Occlusion: Should Emergency Medical Services Transport to the Nearest Primary Stroke Center or Bypass to a Comprehensive Stroke Center With Endovascular Capabilities? Stroke. 2016 Jul;47(7):1965-7. doi: 10.1161/STROKEAHA.115.011149. Epub 2016 Feb 19. No abstract available. PMID 26896433
- [Background] Goyal M, Menon BK, van Zwam WH, Dippel DW, Mitchell PJ, Demchuk AM, Davalos A, Majoie CB, van der Lugt A, de Miquel MA, Donnan GA, Roos YB, Bonafe A, Jahan R, Diener HC, van den Berg LA, Levy EI, Berkhemer OA, Pereira VM, Rempel J, Millan M, Davis SM, Roy D, Thornton J, Roman LS, Ribo M, Beumer D, Stouch B, Brown S, Campbell BC, van Oostenbrugge RJ, Saver JL, Hill MD, Jovin TG; HERMES collaborators. Endovascular thrombectomy after large-vessel ischaemic stroke: a meta-analysis of individual patient data from five randomised trials. Lancet. 2016 Apr 23;387(10029):1723-31. doi: 10.1016/S0140-6736(16)00163-X. Epub 2016 Feb 18. PMID 26898852
- [Background] Jovin TG, Chamorro A, Cobo E, de Miquel MA, Molina CA, Rovira A, San Roman L, Serena J, Abilleira S, Ribo M, Millan M, Urra X, Cardona P, Lopez-Cancio E, Tomasello A, Castano C, Blasco J, Aja L, Dorado L, Quesada H, Rubiera M, Hernandez-Perez M, Goyal M, Demchuk AM, von Kummer R, Gallofre M, Davalos A; REVASCAT Trial Investigators. Thrombectomy within 8 hours after symptom onset in ischemic stroke. N Engl J Med. 2015 Jun 11;372(24):2296-306. doi: 10.1056/NEJMoa1503780. Epub 2015 Apr 17. PMID 25882510
- [Background] Hastrup S, Damgaard D, Johnsen SP, Andersen G. Prehospital Acute Stroke Severity Scale to Predict Large Artery Occlusion: Design and Comparison With Other Scales. Stroke. 2016 Jul;47(7):1772-6. doi: 10.1161/STROKEAHA.115.012482. Epub 2016 Jun 7. PMID 27272487
- [Derived] Behrndtz A, Blauenfeldt RA, Johnsen SP, Valentin JB, Gude MF, Al-Jazi MA, von Weitzel-Mudersbach P, Modrau B, Damgaard D, Hougaard KD, Hjort N, Diedrichsen T, Poulsen M, Schmitz ML, Fisher M, Andersen G, Simonsen CZ; TRIAGE-STROKE Trial Investigators. Transport Strategy in Patients With Suspected Acute Large Vessel Occlusion Stroke: TRIAGE-STROKE, a Randomized Clinical Trial. Stroke. 2023 Nov;54(11):2714-2723. doi: 10.1161/STROKEAHA.123.043875. Epub 2023 Oct 6. PMID 37800374
- See also: national clinical guidelines — http://neuro.dk/wordpress/nnbv/om-iskaemisk-apopleksi/
- See also: Danish Stroke Registry — https://www.rkkp.dk/kvalitetsdatabaser/databaser/dansk-apopleksiregister/